CLINICAL TRIAL: NCT03516851
Title: Multimodal Neuronavigation Guiding Precision Bypass in Adult Ischemic Patients With Moyamoya Disease
Brief Title: Precision Bypass in Patients With Moyamoya Disease
Acronym: PBM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: there are not enough participants enrolled
Sponsor: Peking University International Hospital (Other)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, yuanli Zhao，, professor, Peking University International Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pkuihsw1
Record Dates: First submitted 2018-04-21; First posted 2018-05-04 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Moyamoya Disease
Keywords: Moyamoya Disease; multimodal neuronavigation; flow800; direct revascularization
MeSH Terms: conditions — Moyamoya Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Precision bypass group (Active Comparator): Using ICG with Flow800 software and multimodal neuronavigation to choose the recipient vessel
  Interventions: Procedure: Precision bypass group
- Empirical group (No Intervention): choosing the recipient vessel by the surgeon's own experience

INTERVENTIONS:
Procedure: Precision bypass group — With the brain cortex exposed after craniotomy, an initial ICG fluorescence angiography will be performed. ICG fluorescence angiography using Flow800 software to determine blood flow velocity and cortical perfusion in different candidate receptors. And electromagnetic neuronavigation system is used to evaluate the cerebral flow under different candidate recipient vessels. The treatment planning station will be situated based on the multimodal neuronavigation data. The vessel was chose as the receptor with lower flow velocity and lower cerebral perfusion area to perform anastomosis. Then a direct bypass surgery will be performed just like in the empirical direct bypass surgery group.
  Arms: Precision bypass group

SUMMARY:
Extracranial-intracranial arterial bypass, including anastomosis of the superficial temporal artery to the middle cerebral artery and indirect bypass, can help prevent further ischaemic attacks in patients with Moyamoya disease (MMD). However, there is no established standard for the selection of the recipient vessels. In most situations, surgeons choose the recipient vessels with their own experiences. Intraoperative Indocyanine green (ICG) angiography using Flow800 software and multimodal neuronavigation can be used to assess the real-time cerebral blood flow velocity and perfusion of local brain tissue for better selection of the recipient vessels. Thus the aim of this study is to to determine whether direct bypass surgery combined with multimodal neuronavigation is superior to traditional direct bypass procedure alone in adult ischemic MMD patients.

DETAILED DESCRIPTION:
There are no effective medical therapies for moyamoya disease. Through the provision of collateral pathways, surgical revascularisation is the most successful therapy to improve cerebral haemodynamics, and to reduce the risk of subsequent stroke. Surgical procedures for moyamoya disease can be classified into three categories: direct bypass, indirect bypass, and combined bypass. Although surgeons have their own experience choosing the recipient vessels,no standard has been established based on a worldwide consensus.

Intraoperative ICG angiography using Flow800 software and multimodal neuronavigation (structure combined with perfusion MRI sequence) can be used to assess the real-time cerebral blood flow velocity and perfusion of local brain tissue, which is contribute to choose a recipient vessels with relative low cerebral blood flow velocity and perfusion.

Therefore,the PBM study in our institution is designed to compare the direct bypass surgery with multimodal neuronavigation with traditional direct bypass procedure alone in preventing any ischemic event afterwards after cerebral revascularization surgery in adult ischemic MMD patients.

ELIGIBILITY:
Inclusion Criteria:

* Independent in activity of daily living(The modified Rankin Scale 0-2)
* At least one month since the most recent ischemic stroke
* The neurological deficit must be stable for more than 6 weeks
* Digital substraction angiography demonstrating progressive stenosis or occlusion in the terminal portion of the internal carotid artery and/or the initial portion of the anterior or middle cerebral arteries
* Digital substraction angiography demonstrating formation of abnormal collateral networks (moyamoya vessels) at the base of the brain, mainly in the region of thalamus and basal ganglia
* Digital substraction angiography demonstrating the vasculopathy appeared unilaterally or bilaterally
* Competent to give informed consent
* Accessible and reliable for follow-up

Exclusion Criteria:

* Other diseases(such as internal carotid artery stenosis, internal carotid artery dissection, atrial fibrillation, or Intracranial atherosclerosis) probably causing ischemic strokes
* Not independent in activity of daily living(The modified Rankin Scale 3-5)
* Moyamoya syndrome concomitant with other hereditary or autoimmune diseases (Grave's Disease,Type I Diabetes Mellitus,Type I Neurofibromatosis et al)
* Patient whose initial onset was marked by ischemia but subsequently suffered from intracranial hemorrhage
* Emergent evacuation of intracerebral hematoma damaging superficial temporal artery or cortical artery
* Emergent decompressive craniotomy causing automatically developed indirect revascularization
* Good collateral networks formed by spontaneous anastomosis between extracranial and intracranial vessels before surgery
* Life expectancy<1 years
* Pregnancy
* Unstable angina or myocardial infarction with recent 6 months
* Blood coagulation dysfunction
* Allergic to iodine contrast agent
* Abnormal liver function(alanine transaminase (ALT) and/or aspartate aminotransferase (AST)>3 times of normal range)
* Serum creatinine >3mg/dl
* Poorly controlled hypertension (systolic BP>160 mmHg,diastolic BP>100 mmHg)
* Poor glucose control (fasting blood glucose>16.7mmol/l)
* Concurrent participation in any other interventional clinical trial
* patients refused to participate in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
ischemic events | 30 days
  All strokes & death within 30 days post-surgery and ipsilateral infarctions afterwards

SECONDARY OUTCOMES:
postoperative complications | 30 days
  All kinds of adverse events related to surgery within 30 days
Infarctions | 1 years
  Infarctions on the contralateral side within 1 year of randomization
Transient ischemic attack (TIA) | 1 years
  Transient ischemic attack on the surgically treated side within 1 year of randomization
Cerebral Blood Flow (CBF) | at 7days, 3 months, 6 months, 12 months or end of trial
  The changes from baseline in CBF measured by arterial spin labeling (ASL) at 7days, 3 months, 6 months, 12 months or end of trial
modified Rankin Scale (mRS) | at 7 days, 3 months, 6 months, 12 months or end of trial
  The changes from baseline in modified Rankin Scale (mRS) at 7 days, 3 months, 6 months, 12 months or end of trial. The mRS ranges from 0-6. A mRS of 0-2 is identified as a favourable outcome, and a score of 3-6 as an unfavourable outcome.
National Institute of Health Stroke Scale (NIHSS) | at 7 days, 3 months, 6 months, 12 months or end of trial
  The changes from baseline in National Institute of Health Stroke Scale (NIHSS) at 7 days, 3 months, 6 months, 12 months or end of trial. A total score will be calculated and ranges from 0-42. A NIHSS of 0-14 is identified as a favourable outcome, and a score of 15-42 as an unfavourable outcome.
modified Barthel Index | at 7 days, 3 months, 6 months, 12 months or end of trial
  The changes from baseline in modified Barthel Index at 7 days, 3 months, 6 months, 12 months or end of trial

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolin Chen, PhD, Study Director — Beijing Tiantan Hospital; Junlin Lu, MD, Study Chair — Beijing Tiantan Hospital
Locations (2):
- China (2):
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University International Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Yes
The study protocol of this study is to be shared
Supporting Information: Study Protocol
Time Frame: from September 1, 2018 to September 1, 2019
Access Criteria: everyone

REFERENCES:
- [Background] Scott RM, Smith ER. Moyamoya disease and moyamoya syndrome. N Engl J Med. 2009 Mar 19;360(12):1226-37. doi: 10.1056/NEJMra0804622. No abstract available. PMID 19297575
- [Background] Kuroda S, Houkin K. Moyamoya disease: current concepts and future perspectives. Lancet Neurol. 2008 Nov;7(11):1056-66. doi: 10.1016/S1474-4422(08)70240-0. PMID 18940695
- [Background] Wakai K, Tamakoshi A, Ikezaki K, Fukui M, Kawamura T, Aoki R, Kojima M, Lin Y, Ohno Y. Epidemiological features of moyamoya disease in Japan: findings from a nationwide survey. Clin Neurol Neurosurg. 1997 Oct;99 Suppl 2:S1-5. doi: 10.1016/s0303-8467(97)00031-0. PMID 9409395
- [Background] Caldarelli M, Di Rocco C, Gaglini P. Surgical treatment of moyamoya disease in pediatric age. J Neurosurg Sci. 2001 Jun;45(2):83-91. PMID 11533532
- [Background] Suzuki J, Kodama N. Moyamoya disease--a review. Stroke. 1983 Jan-Feb;14(1):104-9. doi: 10.1161/01.str.14.1.104. PMID 6823678
- [Background] Baba T, Houkin K, Kuroda S. Novel epidemiological features of moyamoya disease. J Neurol Neurosurg Psychiatry. 2008 Aug;79(8):900-4. doi: 10.1136/jnnp.2007.130666. Epub 2007 Dec 12. PMID 18077479
- [Derived] Lu J, Zhao Y, Ma L, Chen Y, Li M, Ye X, Wang R, Chen X, Zhao Y. Multimodal neuronavigation-guided precision bypass in adult ischaemic patients with moyamoya disease: study protocol for a randomised controlled trial. BMJ Open. 2019 Mar 20;9(3):e025566. doi: 10.1136/bmjopen-2018-025566. PMID 30898819